CLINICAL TRIAL: NCT01130857
Title: Diagnostic Tools in Temporal Arteritis - Towards the Development of a Diagnostic Algorithm
Brief Title: Diagnostic Study of Temporal Arteritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Israel Heller MD, Israel Heller MD, Tel-Aviv Sourasky Medical Center
Other Study IDs: 0123-09-TLV
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-01

CONDITIONS: Temporal Arteritis
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite a large and growing body of knowledge concerning the diagnosis of temporal arteritis, this potentially crippling disease still requires pathological diagnosis in practically every case. It seems likely that a correctly estimated clinical probability could help in evaluating imaging results in a way that might safely obviate temporal biopsy in a large segment of suspect cases.

With this aim in view, we intend to identify useful clinical items and integrate them in an appropriate diagnostic pathway.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of temporal arteritis and referred by their physicians to biopsy of a temporal artery.

Exclusion Criteria:

* Pregnancy; age > 80 or < 18; unable to answer study questions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients suspected of temporal arteritis and referred to temporal artery biopsy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-03 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Percent decrease in future biopsy use. | 2 years

SECONDARY OUTCOMES:
No secondary outcome. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Israel SA Heller, MD, Principal Investigator — Tel Aviv Medical Center, Tel Aviv, ISRAEL